CLINICAL TRIAL: NCT01934660
Title: Inflammatory Characterization of Known or Possible Cardiovascular Diseases
Brief Title: Links Between Inflammation and Cardiometabolic Diseases
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 130194; 13-H-0194
Record Dates: First submitted 2013-08-28; First posted 2013-09-04 (Estimated); Last update posted 2025-12-31 (Actual); Status verified 2025-09-22

CONDITIONS: Diabetes Mellitus; Cardiovascular Disease; Healthy Volunteer; Inflammation
Keywords: Cardiovascular Disease; Diabetes Mellitus; Inflammation; Natural History
MeSH Terms: conditions — Diabetes Mellitus; Cardiovascular Diseases; Inflammation | interventions — Fluorodeoxyglucose F18

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: Healthy volunteers
  Interventions: Drug: 13N-amonia; Drug: Fludeoxyglucose F18
- Group 2: Subjects diagnosed with diabetes
  Interventions: Drug: 13N-amonia; Drug: Fludeoxyglucose F18
- Group 3: Subjects diagnosed cardiovascular disease
  Interventions: Drug: 13N-amonia; Drug: Fludeoxyglucose F18

INTERVENTIONS:
Drug: 13N-amonia — PET/Scan
Drug: Fludeoxyglucose F18 — PET/Scan

SUMMARY:
Background:

- Cardiometabolic diseases are a combination of medical disorders that, when they occur together, increase the risk of heart disease and diabetes. Researchers want to learn if there is a relationship between these diseases and inflammation (redness, swelling, and pain). Inflammation affects the entire body. Researchers will study this relationship in people with heart disease and diabetes, and compare it to healthy people.

Objectives:

- To learn if there are links between inflammation and cardiometabolic diseases.

Eligibility:

* Adults 18 years of age or older with heart disease or diabetes.
* Healthy volunteers 18 years of age or older.

Design:

* Participants will have up to six study visits. There will be first visit, then an optional visit 12 months after the first visit.
* At the study visits they will have:

  * Blood taken with a needle in their arm.
  * An electrocardiogram. Small patches are stuck to the chest and limbs. A machine measures electrical signals of the heart.
  * Completed a number of questionnaires.
  * A body scan called an FDG PET/CT. A substance will be injected through a tube in their arm. They will lie on a special bed that will move in and out of the PET/CT scanner. The PET/CT scanner will take pictures of the body. The scan will last up to 30 minutes.
  * Some participants will have other body scans ( FDG PET/MRI). The procedures are similar to the FDG PET/CT scan. These other scans will last about 30 minutes total.
  * Some participants will also have a CT scan of their heart. A substance will be injected through a tube in their arm. They will lie on a table in a large, donut-shaped machine. An X-ray tube will move around their body, taking many pictures. This procedure can last up to 2 hours.
  * Some participants will have tests that measures blood pressure and how the blood moves through the body.
  * Some participants will have small samples of skin and fat tissue taken.

DETAILED DESCRIPTION:
Over the past two decades, the number of subjects with cardiometabolic diseases (CMD) such as atherosclerotic cardiovascular disease (CVD), dyslipidemia, insulin resistance and diabetes have been rising. Characterizing these disease states reveals that inflammation is a common feature of CMD; however, mechanistic links between inflammation and these disease states in humans remain poorly understood. In this protocol, we aim to characterize inflammation within the blood vessels, blood, fat and skin in diabetes and coronary artery disease compared to those without disease. We hypothesize that diabetes and coronary disease will be systemic inflammatory states and will provide an important frame of reference for parameters found on novel imaging techniques in another ongoing protocol trying to understand how skin inflammation affects risk for CMD and CVD (13-H-0065).

ELIGIBILITY:
* Cardiovascular Disease Eligibility Criteria

INCLUSION CRITERIA:

* Females and males 18 years of age or older
* Diagnosis of clinical CAD (including abnormal EKG with a prior infarction pattern, abnormal echo consistent with a wall motion abnormality or a referral note from cardiologist with diagnosis of CAD)
* CAD that is currently stable (defined by no change in medications for blood pressure, angina or diuretic therapy or in no new CV symptoms over the past month in a patient who has had a primary cardiac event or an abnormal EKG with confirmed wall motion abnormality)
* CAD which may be associated with chronic stable angina (defined by a clinical syndrome characterized by discomfort in the chest, jaw, shoulder, back, or arm by a physician).
* CAD that is found on CCTA which may be subclinical

EXCLUSION CRITERIA:

* Pregnant women or lactating women.
* For optional adipose biopsy, any subject with known bleeding disorder, current fever or on anti-coagulation.
* For optional MRI, inability to participate due to metal within body, claustrophobia, or anything else that prohibits undergoing a MRI scan
* Any solid organ or liquid tumor within the past five years, with the exception of nonmelanomatous skin cancer,
* Active infectious diseases within 3 months requiring antibiotics, collagen vascular diseases such as RA, psoriasis and mixed connective tissue diseases and immune-mediated lung diseases (e.g. IPF, BOOP)
* A BMI >40 kg/m(2) due to PET MRI restrictions
* Subjects with severe renal excretory dysfunction, estimated glomerular filtration rate < 30 mL/min/1.73m(2) body surface area according to the Modification of Diet in Renal Disease criteria, will not receive the cardiac CT angiography, or gadolinium contrast agent during the PET/MRI.

Diabetes Mellitus Eligibility Criteria

INCLUSION CRITERIA:

* Females and males 18 years of age or older
* Diagnosis of type 2 diabetes mellitus (DM), currently stable as defined by no change in antidiabetic medications over the past month and fasting glucose <200

EXCLUSION CRITERIA:

* Pregnant women and or lactating women.
* For optional adipose biopsy, any subject with known bleeding disorder, current fever or on anti-coagulation.
* For optional MRI, inability to participate due to metal within body, claustrophobia, or anything else that prohibits undergoing a MRI scan
* Any solid organ or liquid tumor within the past five years, with the exception of nonmelanomatous skin cancer,
* Active infectious diseases within 3 months requiring antibiotics, collagen vascular diseases such as RA, psoriasis and mixed connective tissue diseases and immune-mediated lung diseases (e.g. IPF, BOOP)
* A BMI >40 kg/m(2) due to PET MRI restrictions
* Subjects with severe renal excretory dysfunction, estimated glomerular filtration rate < 30 mL/min/1.73m(2) body surface area according to the Modification of Diet in Renal Disease criteria, will not receive the cardiac CT angiography, or gadolinium contrast agent during the PET/MRI.
* Subjects with second -or third-degree AV block or sinus node dysfunction will not receive the 13N-ammonia PET/CT imaging unless these patients have a functioning artificial pacemaker.
* Subjects with any signs or symptoms of acute coronary syndrome, including vasoreactive hypertension with blood pressure exceeding 180/100, any concerning ST segment changes on ECG, or acute chest pain, will not receive the 13N-ammonia PET/CT imaging.

Healthy Volunteers:

INCLUSION CRITERIA:

-Females and males 18 years of age or older without any clinical diagnosis of a chronic health condition that is knownto accelerate vascular disease beyond traditional risk factors including lung disease or active infection

EXCLUSION CRITERIA:

* For imaging studies, pregnant women
* For imaging studies, lactating women
* For optional MRI, inability to participate due to in optional MRI metal within body, claustrophobia, or anything else that prohibits undergoing a MRI scan
* Any solid organ or liquid tumor within the past five years, with the exception of non melanomatous skin cancer,
* Active infectious diseases within 3 months requiring antibiotics, collagen vascular diseases such as RA, psoriasis and mixed connective tissue diseases and immune-mediated lung diseases (e.g. IPF, BOOP)
* Clinical diagnosis of diabetes or cardiovascular disease
* Fasting glucose >125,
* LDL>200,
* LFT s 3 times normal limit,
* eGFR<60,
* Subjects with severe renal excretory dysfunction will not receive the cardiac CT angiography, or gadolinium contrast agent during the PET/MRI.
* A BMI >40 kg/m(2) due to PET MRI restrictions.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers and participants diagnosed with diabetes or cardiovascular disease will be recruited for this protocol.@@@
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2013-12-02 (Actual); Primary Completion 2022-08-03 (Actual)

PRIMARY OUTCOMES:
Our primary outcome of interest is vascular inflammation measured by standard uptake values from PET/CT and PET/MRI imaging with FDG | 1 day to 10 years
  vascular inflammation measured by standard uptake values from PET/CT and PET/MRI imaging with FDG

SECONDARY OUTCOMES:
Our secondary outcomes are mean aortic wall thickness at the most diseased segment on FDG PET/CT and vessel wall area on MRI at the most diseased segment, and we will perform analyses using a model including the same variables as above. | 1 day to 10 years
  Mean Aortic Wall Thickness at the most diseased segment (measured by MRI at FDG PET MRI) --Vessel Wall Area at the most diseased segment (measured by MRI at FDG PET MRI)
As a tertiary analysis, we will add novel biomarkers to the above models including HDL efflux, HOMA-IR and inflammatory mediators to understand the association of each biomarker on vascular disease markers | 1 day to 10 years
  to understand the association of each biomarker on vascular disease markers

CONTACTS AND LOCATIONS:
Overall Officials: Michael N Sack, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Han K, Singh K, Meadows AM, Sharma R, Hassanzadeh S, Wu J, Goss-Holmes H, Huffstutler RD, Teague HL, Mehta NN, Griffin JL, Tian R, Traba J, Sack MN. Boosting NAD preferentially blunts Th17 inflammation via arginine biosynthesis and redox control in healthy and psoriasis subjects. Cell Rep Med. 2023 Sep 19;4(9):101157. doi: 10.1016/j.xcrm.2023.101157. Epub 2023 Aug 15. PMID 37586364
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2013-H-0194.html